CLINICAL TRIAL: NCT05327296
Title: A Phase 3, Multicenter, Randomized, Controlled, Open Label, Assessor-Blinded Study to Evaluate the Efficacy and Safety of Inhaled Isoflurane Delivered Via the Sedaconda ACD-S Compared to Intravenous Propofol for Sedation of Mechanically Ventilated Intensive Care Unit Adult Patients (INSPiRE-ICU2)
Brief Title: Efficacy and Safety of Inhaled Isoflurane Delivered Via the Sedaconda ACD-S Compared to Intravenous Propofol for Sedation of Mechanically Ventilated Intensive Care Unit Adult Patients (INSPiRE-ICU2)
Acronym: INSPiRE-ICU2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sedana Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SED004
Record Dates: First submitted 2022-04-05; First posted 2022-04-14 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Sedation
Keywords: sedation; mechanical ventilation; propofol; ICU; isoflurane
MeSH Terms: interventions — Isoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isoflurane (Experimental): Inhaled isoflurane administered via Sedaconda ACD-S
  Interventions: Drug: Isoflurane
- Propofol (Active Comparator): Propofol administered as intravenous infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Isoflurane — Inhaled isoflurane administered by Sedaconda ACD-S
  Arms: Isoflurane
Drug: Propofol — Intravenous infusion of propofol
  Arms: Propofol

SUMMARY:
This is a study to compare safety and efficacy of inhaled isoflurane administered via the Sedaconda ACD-S device system versus intravenous propofol for sedation of mechanically ventilated patients in the Intensive Care Unit (ICU) setting.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, controlled, open-label, assessor-blinded study to evaluate the efficacy and safety of inhaled isoflurane delivered via the Sedaconda ACD-S compared to intravenous propofol for sedation of mechanically ventilated Intensive Care Unit (ICU) adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age;
* Patients who are anticipated to require >12 hours of invasive mechanical ventilation and continuous sedation in the ICU; and
* Receipt of continuous sedation due to clinical need for sedation to RASS <0.

Exclusion Criteria:

* Need for RASS -5;
* Sedation for invasive mechanical ventilation immediately prior to Baseline for >72 hours;
* Severe neurological condition before ICU admission that causes the patient to lack ability to participate in the study (ie, unable to be assessed for RASS and CPOT);
* Ventilator tidal volume <200 or >1000 mL at Baseline;
* Need for extracorporeal membrane oxygenation (ECMO), extracorporeal CO2 removal (ECCO2R), high frequency oscillation ventilation (HFOV), or high frequency percussive ventilation (HFPV) at Screening;
* Comfort care only (end of life care);
* Contraindication to propofol or isoflurane;
* Known or family history of MH;
* Severe hemodynamic compromise, defined as the need for norepinephrine ≥0.3 mcg/kg/min (or equivalent vasopressor dose) to maintain blood pressure within acceptable range, assumed to be mean arterial pressure ≥65 mmHg unless prescribed clinically;
* Allergy to isoflurane or propofol, or have propofol infusion syndrome.
* History of ventricular tachycardia/Long QT Syndrome;
* Requirement of IV benzodiazepine or barbiturate administration for seizures or dependencies, including alcohol withdrawal
* Neuromuscular disease that impairs spontaneous ventilation (eg, C5 or higher spinal cord injury, amyotrophic lateral sclerosis, etc);
* Concurrent enrollment in another study that, in the Investigator's opinion, would impact the patient's safety or assessments of this study;
* Participation in other study involving investigational drug(s) or devices(s) within 30 days prior to Randomization;
* Anticipated requirement of treatment with continuous infusion of a neuromuscular blocking agent for >4 hours;
* Female patients who are pregnant or breast-feeding;
* Imperative need for continuous active humidification through mechanical ventilation circuit;
* Attending physician's refusal to include the patient; or
* Inability to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of time adequate sedation depth | During study treatment up to 48 (±6) hours
  To compare the percentage of time sedation depth is maintained within the target range, in absence of rescue sedation, as assessed according to the RASS scale, in isoflurane- vs propofol-treated patients

SECONDARY OUTCOMES:
Key Secondary: Compare the use of opioids | During study treatment up to 48 (±6) hours
  To compare the effect of isoflurane vs propofol on use of opioids during the study drug treatment period measuring CPOT
Key Secondary: Compare the wake up time | Time from stop of study drug treatment up to 4 hours
  To compare the effect of isoflurane vs propofol on the wake up time at end of study drug treatment
Key Secondary: Compare the cognitive recovery after EOT | 60 minutes after EOT
  To compare the effect of isoflurane vs propofol on cognitive recovery after EOT by measuring CAM-ICU-7
Key Secondary: Compare the spontaneous breathing effort | During study treatment up to 48 (±6) hours
  To compare the effect of isoflurane vs propofol on spontaneous breathing effort during the study drug treatment period by measuring
  • Airway occlusion pressure, pressure support or if observed respiratory rate exceeds set respiratory rate
Other secondary: Compare time from sedation termination to extubation | During study treatment
  To compare the effect of isoflurane vs propofol on time from sedation termination to extubation in patients for whom study drug is terminated for extubation
Other secondary: Compare days alive and free of mechanical ventilation through Study Day 30 | From start of study treatment up to 30 days
  To compare the effect of isoflurane vs propofol on days alive and free of mechanical ventilation through Study Day 30
Other secondary: Compare days alive and free of the ICU | From start of study treatment up to 30 days
  To compare the effect of isoflurane vs propofol on days alive and free of the ICU
Other secondary: Compare delirium and coma free days until 7 days after EOT | From start of study treatment until 7 days after EOT
  To compare the effect of isoflurane vs propofol on delirium and coma free days until 7 days after EOT
Other secondary: Compare mortality at 30 days after randomization | Until 30 days after randomization
  To compare the effect of isoflurane vs propofol on mortality at 30 days after randomization
Other secondary: Compare mortality at 3 months after randomization | Until 3 months after randomization
  To compare the effect of isoflurane vs propofol on mortality at 3 months after randomization
Other secondary: Compare mortality at 6 months after randomization | Until 6 months after randomization
  To compare the effect of isoflurane vs propofol on mortality at 6 months after randomization
Other secondary: To compare the safety profile of isoflurane vs propofol | Baseline to end of study treatment, safety lab from baseline up to 48hrs post treatment, AEs from start study treatment up to day 30
  To compare the safety profile of isoflurane vs propofol in respect to reported Adverse Event
Other secondary: To assess Sedaconda ACD-S device deficiencies in patients receiving isoflurane | During study treatment up to 48 (±6) hours
  To assess Sedaconda ACD-S device deficiencies in patients receiving isoflurane by Sedaconda ACD-S by reported Adverse Event
Other secondary: To compare the use of restraints in patients receiving isoflurane vs propofol | During study treatment up to 48 (±6) hours
  Incidence of restraints measured twice daily

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Beitler, M.D., Principal Investigator — Columbia University
Locations (16):
- United States (16):
  - Memorial Health Services, Long Beach, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - University of California, San Diego, San Diego, California
  - University of Miami, Coral Gables, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - The Cooper Health System, Camden, New Jersey
  - The New York and Presbyterian Hospital, New York, New York
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Memorial Hermann Health Services, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Shehabi Y, Howe BD, Bellomo R, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Murray L, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; ANZICS Clinical Trials Group and the SPICE III Investigators. Early Sedation with Dexmedetomidine in Critically Ill Patients. N Engl J Med. 2019 Jun 27;380(26):2506-2517. doi: 10.1056/NEJMoa1904710. Epub 2019 May 19. PMID 31112380
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503
- [Background] Sackey PV, Martling CR, Carlsward C, Sundin O, Radell PJ. Short- and long-term follow-up of intensive care unit patients after sedation with isoflurane and midazolam--a pilot study. Crit Care Med. 2008 Mar;36(3):801-6. doi: 10.1097/CCM.0B013E3181652FEE. PMID 18431266
- [Background] Mesnil M, Capdevila X, Bringuier S, Trine PO, Falquet Y, Charbit J, Roustan JP, Chanques G, Jaber S. Long-term sedation in intensive care unit: a randomized comparison between inhaled sevoflurane and intravenous propofol or midazolam. Intensive Care Med. 2011 Jun;37(6):933-41. doi: 10.1007/s00134-011-2187-3. Epub 2011 Mar 29. PMID 21445642
- [Background] Meiser A, Volk T, Wallenborn J, Guenther U, Becher T, Bracht H, Schwarzkopf K, Knafelj R, Faltlhauser A, Thal SC, Soukup J, Kellner P, Druner M, Vogelsang H, Bellgardt M, Sackey P; Sedaconda study group. Inhaled isoflurane via the anaesthetic conserving device versus propofol for sedation of invasively ventilated patients in intensive care units in Germany and Slovenia: an open-label, phase 3, randomised controlled, non-inferiority trial. Lancet Respir Med. 2021 Nov;9(11):1231-1240. doi: 10.1016/S2213-2600(21)00323-4. Epub 2021 Aug 26. PMID 34454654
- [Background] Kong KL, Willatts SM, Prys-Roberts C. Isoflurane compared with midazolam for sedation in the intensive care unit. BMJ. 1989 May 13;298(6683):1277-80. doi: 10.1136/bmj.298.6683.1277. PMID 2500195
- [Background] Chanques G, Constantin JM, Devlin JW, Ely EW, Fraser GL, Gelinas C, Girard TD, Guerin C, Jabaudon M, Jaber S, Mehta S, Langer T, Murray MJ, Pandharipande P, Patel B, Payen JF, Puntillo K, Rochwerg B, Shehabi Y, Strom T, Olsen HT, Kress JP. Analgesia and sedation in patients with ARDS. Intensive Care Med. 2020 Dec;46(12):2342-2356. doi: 10.1007/s00134-020-06307-9. Epub 2020 Nov 10. PMID 33170331
- [Background] Jerath A, Ferguson ND, Cuthbertson B. Inhalational volatile-based sedation for COVID-19 pneumonia and ARDS. Intensive Care Med. 2020 Aug;46(8):1563-1566. doi: 10.1007/s00134-020-06154-8. Epub 2020 Jun 25. PMID 32588067
- [Background] Bellgardt M, Bomberg H, Herzog-Niescery J, Dasch B, Vogelsang H, Weber TP, Steinfort C, Uhl W, Wagenpfeil S, Volk T, Meiser A. Survival after long-term isoflurane sedation as opposed to intravenous sedation in critically ill surgical patients: Retrospective analysis. Eur J Anaesthesiol. 2016 Jan;33(1):6-13. doi: 10.1097/EJA.0000000000000252. PMID 25793760
- [Background] Hughes CG, Mailloux PT, Devlin JW, Swan JT, Sanders RD, Anzueto A, Jackson JC, Hoskins AS, Pun BT, Orun OM, Raman R, Stollings JL, Kiehl AL, Duprey MS, Bui LN, O'Neal HR Jr, Snyder A, Gropper MA, Guntupalli KK, Stashenko GJ, Patel MB, Brummel NE, Girard TD, Dittus RS, Bernard GR, Ely EW, Pandharipande PP; MENDS2 Study Investigators. Dexmedetomidine or Propofol for Sedation in Mechanically Ventilated Adults with Sepsis. N Engl J Med. 2021 Apr 15;384(15):1424-1436. doi: 10.1056/NEJMoa2024922. Epub 2021 Feb 2. PMID 33528922
- [Background] Krannich A, Leithner C, Engels M, Nee J, Petzinka V, Schroder T, Jorres A, Kruse J, Storm C. Isoflurane Sedation on the ICU in Cardiac Arrest Patients Treated With Targeted Temperature Management: An Observational Propensity-Matched Study. Crit Care Med. 2017 Apr;45(4):e384-e390. doi: 10.1097/CCM.0000000000002185. PMID 27941501
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Derived] O'Gara B, Serra AL, Englert JA, Sachdev A, Owens RL, Chang SY, Park PK, Talmor D, Sverud I, Sackey P, Beitler JR. Inhaled sedation versus propofol in respiratory failure in the ICU (INSPiRE-ICU2): study protocol for a multicenter randomized controlled trial. Trials. 2025 Mar 31;26(1):114. doi: 10.1186/s13063-025-08791-0. PMID 40165305
- See also: Isoflurane 100% inhalation vapour, liquid. Summary of product characteristics. West Drayton, United Kingdon. Piramal Critical Care Ltd. Electronic medicines compendium(emc), last updated 29 October 2019. Accessed 09 September 2020. — http://www.medicines.org.uk/emc/product/9800/smpc#gref